CLINICAL TRIAL: NCT01435928
Title: A Double-Blind, Placebo-Controlled, Randomized Withdrawal Study Of Lurasidone For The Maintenance Treatment Of Subjects With Schizophrenia
Brief Title: PEARL Schizophrenia Maintenance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1050238
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Lurasidone; Latuda
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lurasidone (Experimental): Lurasidone 40 and 80 mg, once daily in the evening with a meal or 30 minutes after eating
  Interventions: Drug: Lurasidone
- Placebo (Placebo Comparator): Matching placebo once daily in the evening with a meal or 30 minutes after eating
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Lurasidone — Lurasidone 40 and 80 mg, once daily in the evening with a meal or 30 minutes after eating
  Other Names: Latuda
  Arms: Lurasidone
Drug: Matching Placebo — Matching placebo once daily in the evening with a meal or 30 minutes after eating
  Arms: Placebo

SUMMARY:
Lurasidone HCI is a compound that is FDA-approved for the treatment of schizophrenia. This clinical study is designed to test the hypothesis that Lurasidone is effective in the long term maintenance treatment of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

Open Label:

Subject provides written informed consent and is willing and able to comply with the protocol in the opinion of the Investigator.

Subject is ≥ 18 and ≤ 75 years of age, on the day of signing the informed consent.

Subject meets DSM-IV-TR criteria for a primary diagnosis of schizophrenia [including disorganized (295.10), paranoid (295.30), undifferentiated (295.90) subtypes as established by clinical interview (using the DSM-IV-TR as a reference and confirmed using the SCID-CT)]. The duration of the subject's illness whether treated or untreated must be ≥ 1 year.

Subject has had at least one prior episode of psychotic exacerbation as judged by the Investigator in the two years preceding screening.

Subject has a PANSS Total score ≥ 80 with a score ≥ 4 on 1 or more of any PANSS Positive subscale items at screening and open-label baseline (Visit 2).

Subject has a CGI-S score of ≥ 4 at screening and open-label baseline (Visit 2).

Subject is not pregnant (must have a negative serum pregnancy test at screening) or nursing (must not be lactating) and is not planning pregnancy within the projected duration of the study.

Female subject of reproductive potential agrees to remain abstinent or use adequate and reliable contraception throughout the study and for at least 30 days after the last dose of lurasidone has been taken. In the Investigator's judgment, the subject will adhere to this requirement.

Adequate contraception is defined as continuous use of either two barrier methods (e.g., condom and spermicide or diaphragm with spermicide) or a hormonal contraceptive. Acceptable hormonal contraceptives include the following: a) contraceptive implant (such as Norplant®) implanted at least 90 days prior to screening; b) injectable contraception (such as medroxyprogesterone acetate injection) given at least 14 days prior to screening; or c) oral contraception taken as directed for at least 30 days prior to screening.

Subjects who are of non-reproductive potential, i.e., subject who is surgically sterile, has undergone tubal ligation, or is postmenopausal (defined as at least 12 months of spontaneous amenorrhea or between 6 and 12 months of spontaneous amenorrhea with follicle stimulating hormone (FSH) concentrations within postmenopausal range as determined by laboratory analysis) are not required to remain abstinent or use adequate contraception.

Subject is able and agrees to remain off prior antipsychotic medication for the duration of the study.

Subject has had a stable living arrangement at the time of screening and agrees to return to a similar living arrangement after discharge, if hospitalized. This criterion is not meant to exclude subjects who have temporarily left a stable living arrangement (e.g., due to psychosis). Such subjects remain eligible to participate in this protocol. Chronically homeless subjects should not be enrolled.

Subject is in good physical health on the basis of medical history, physical examination, and laboratory screening.

Subject who requires concomitant medication treatment with the following agents may be included if they have been on stable doses (i.e., minor adjustments only) for the specified times: 1) antidepressant agents (except fluvoxamine) and/or mood stabilizers (except carbamazepine or oxcarbazepine) must be stable for at least 30 days prior to open-label baseline, 2) oral hypoglycemics must be stable for at least 30 days prior to screening, 3) antihypertensive agents must be stable for at least 30 days prior to screening, and 4) thyroid hormone replacement must be stable for at least 90 days prior to screening. (Note: CYP3A4 inducers and inhibitors will not be allowed).

Subject is willing and able to comply with the protocol assessments and visits, in the opinion of the study nurse/coordinator and the Investigator.

Double-blind -

Subject must achieve and maintain clinical stability for a total of at least 12 weeks in the open label phase, defined as:

1. a PANSS Total score ≤ 70, a CGI-S score < 4 and a PANSS item score of ≤ 4 (moderate or less) on all PANSS Positive subscale items over at least 12 weeks with the allowance of two excursions (except during the last 4 weeks of the open-label phase) assessed at weekly study visits:

   • An excursion is defined as a PANSS total score up to a maximum of 80 and/or a CGI-S score up to a maximum of 4 and/or a PANSS Positive subscale item score up to a maximum of 5.
2. a PANSS item score of ≤ 4 (moderate or less) on item G8 (uncooperativeness)
3. taking a stable dose of lurasidone for the last 4 weeks of the open-label phase.

Exclusion Criteria:

Open Label - Subject has a DSM-IV Axis I or Axis II diagnosis other than schizophrenia that has been the primary focus of treatment within 3 months of screening.

Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at screening (in the past month) or baseline.

Subject has attempted suicide within 3 months prior to the screening phase. Subject currently has a clinically significant medical condition including the following: neurological, metabolic (including Type 1 diabetes), hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, and/or urological disorder such as unstable angina, congestive heart failure (uncontrolled), or central nervous system (CNS) infection that would pose a risk to the subject if they were to participate in the study or that might confound the results of the study. Subjects with human immunodeficiency virus (HIV) seropositivity (or history of seropositivity) will be excluded.

Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Monitor should be consulted. Any subject with a known cardiovascular disease or condition (even if controlled) must be discussed with the Medical Monitor before being screened.

Subject has evidence of any chronic organic disease of the CNS such as tumors, inflammation, and active seizure disorder, vascular disorder, Parkinson's disease, Alzheimer's disease or other forms of dementia, myasthenia gravis, or other degenerative processes. In addition, subject must not have a history of mental retardation or persistent neurological symptoms attributable to serious head injury. Note: Past history of febrile seizures, drug-induced seizures, or alcohol withdrawal seizures is not exclusionary.

Note: Past history of febrile seizures, drug-induced seizures, or alcohol withdrawal seizures is not exclusionary.

Subject demonstrates evidence of acute hepatitis, clinically significant chronic hepatitis, or evidence of clinically significant impaired hepatic function through clinical and laboratory evaluation.

Note: Subjects with serum alanine transaminase (ALT) or aspartate transaminase (AST) levels ≥ 3 times the upper limit of the reference ranges provided by the central laboratory require retesting. If on retesting, the laboratory value remains ≥ 3 times the upper limit, such subjects will be discussed with the Medical Monitor for enrollment consideration.

Subject has a history of stomach or intestinal surgery or any other condition that could interfere with or is judged by the Investigator to interfere with absorption, distribution, metabolism, or excretion of study drug.

Subject with Type 1 or Type 2 insulin-dependent diabetes.

Subject with newly diagnosed Type 2 diabetes during screening. Subject with Type 2 diabetes is eligible for study inclusion if the following condition is met at screening:

if a subject is currently being treated with oral anti-diabetic medication(s), the dose must have been stable for at least 4 weeks prior to screening. Such medication may be adjusted or discontinued during the study, as clinically indicated.

Subject has any abnormal laboratory parameter at screening that indicates a clinically significant medical condition as determined by the Investigator. Subjects with a fasting blood glucose at screening ≥ 126 mg/dL (7.0 mmol/L) or HbA1c ≥ 7.0% will be excluded.

Note: Subjects with random (non-fasting) blood glucose at screening ≥ 200 mg/dL (11.1 mmol/L) must be retested in a fasted state.

Subject has a prolactin concentration > 100 ng/mL at screening or has a history of pituitary adenoma.

Subject has a history of malignancy < 5 years prior to signing the informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Pituitary tumors of any duration are excluded.

Subject is judged to be resistant to antipsychotic treatment defined as any one of the following:

1. failure to respond to > 2 marketed antipsychotic agents, given at an adequate dose and for an adequate duration (within the past 2 years)
2. history of treatment with clozapine for refractory psychosis Subject is unlikely to achieve a stable condition for ≥ 12 weeks during the open-label lurasidone phase based on the totality of evidence from the psychiatric history and/or the current presentation.

Subject is receiving an antipsychotic medication above the maximum recommended (country-specific) dose at or prior to screening and, in the judgment of the Investigator, is unlikely to respond to standard doses of lurasidone.

Subject has received depot antipsychotics unless the last injection was at least one treatment cycle or at least 30 days (whichever is longer) prior to the screening phase.

Subject has received treatment with MAO inhibitors within 14 days prior to the screening phase.

Subject requires treatment with any potent CYP3A4 inhibitors or inducers during the study (see Appendix 3).

Subject has received electroconvulsive therapy treatment within the 3 months prior to screening or is expected to require electroconvulsive therapy (ECT) during the study.

Subject has a history of neuroleptic malignant syndrome. Subject exhibits evidence of severe tardive dyskinesia, severe dystonia, or any other severe movement disorder. Severity will be determined by the Investigator.

Subject has a history of alcohol or substance abuse (DSM-IV-TR criteria) within 3 months prior to screening or alcohol or substance dependence (DSM-IV-TR criteria) within 12 months prior to screening. The only exceptions include caffeine or nicotine abuse/dependence.

Subject tests positive for drugs of abuse at screening. In the event a subject tests positive for cannabinoids (tetrahydrocannabinol), the Investigator will evaluate the subject's ability to abstain from using this drug during the study. This information will be discussed with the Medical Monitor prior to study enrollment.

Subject had a history or presence of an abnormal electrocardiogram (ECG), which in the Investigator's opinion is clinically significant (Medical Monitor may be consulted to determine clinical significance).

Subject has poor peripheral venous access that will limit the ability to draw blood as judged by the Investigator.

Subject has a history of hypersensitivity to more than 2 distinct chemical classes of drug (e.g., sulfas and penicillins).

Subject was screened or washed out previously more than three times for this study.

Subject is currently participating, or has participated in, a study with an investigational or marketed compound or device within 3 months prior to signing the informed consent, or has participated in 2 or more studies within 12 months prior to signing the informed consent.

Subject is homeless or did not have a stable residence for the 3 months prior to the screening phase.

Subject is unable to cooperate with any study procedures, unlikely to adhere to the study procedures and keep appointments, in the opinion of the Investigator, or was planning to relocate during the study.

Subject requires guardianship under the laws of his/her country.

Double-blind - Subjects who in the Investigator's judgment have not been compliant with study medication during the open-label stabilization phase.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (75):
- United States (45):
  - Woodland Research Northwest, Springdale, Arizona
  - K&S Professional Research, Little Rock, Arkansas
  - Woodland International Research Group, Little Rock, Arkansas
  - Comprehensive Clinical Development Inc., Cerritos, California
  - Diligent Clinical Trials, Downey, California
  - Synergy Escondido, Escondido, California
  - Collaborative Neuroscience Network, Inc., Garden Grove, California
  - Axis Clinical Trials, Los Angeles, California
  - Synergy Clinical Research Center, National City, California
  - Excell Clinical Trials, Oceanside, California
  - CNRI - Los Angeles LLC,8309 Telegraph Road, Pico Rivera, California
  - California Neuropsychopharmacology Clinical Research Instit, San Diego, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Collaborative Neuroscience Network Inc., Torrance, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Accurate Clinical Trials, Kissimme, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Galiz Research, Miami Springs, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Comprehensive NeuroScience, Inc., Atlanta, Georgia
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Lousiana Clinical Research, LLC, Shreveport, Louisiana
  - CBH Health LLC, Rockville, Maryland
  - Psychiatric Care and Research Center, O'Fallon, Missouri
  - Psych Care Consultants Research, St Louis, Missouri
  - Horne Research, Las Vegas, Nevada
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - CRI Worldwide LLC, Willingboro, New Jersey
  - University of New York, Dept. of Psychiatry, Buffalo, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Comprehensive Clinical Development, Inc, Fresh Meadows, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Oklahoma Clinical Research, Oklahoma City, Oklahoma
  - CRI Worldwide LLC at Kirkbride, Philadelphia, Pennsylvania
  - Lincoln Research, Lincoln, Rhode Island
  - Community Clinical Research, Inc., Austin, Texas
  - FutureSearch Clinical Trials LP, Austin, Texas
  - FutureSearch Clinical Trials, LP, Dallas, Texas
  - Pillar Clinical Research LLC, Dallas, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Department of Psychiatry, University of Utah Health Sciences Center, Salt Lake City, Utah
  - Frontier Institute, Spokane, Washington
- France (5):
  - CHU Clermont-Ferrand - CMP B, Clermont-Ferrand
  - Centre Hospitalier Specialise du Jura - Centre Medico Psychiatric, Dole
  - Centre Hospitalier Guillaume Regnier, Rennes
  - Hopital Chalucet, Centre hospitalier intercommunal de toulon la Seyne sur mer (CHITS), Toulon
  - Cabinet Medical, Toulouse
- Italy (3):
  - SC SPDC-Edificio n. 7, Ospedale S. Andrea, La Spezia
  - Dipartimento Salute Mentale ASL 1, Massa
  - A.O.U. Santa Chiara, U.O di Psichiatria 1 building n.4, Pisa
- Russia (6):
  - Regional Government Institution Kipetsk Regional Psychoneurology Hospital, Lipetsk
  - Limited Liability Company (LLC) Research Center for Treatment and rehabilitation "Phoenix", Rostov-on-Don
  - City Psychoneurological Dispensary #7 (with Hospital), Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution City Psychoneurology Dispensary #7 (with in-patient dept.) (SPb SBHI CPNDD-7), at daycare facility #1, Saint Petersburg
  - St. Petersburg State Healthcare Institution (SPbSH) "City Psychiatric Hospital #6", Saint Petersburg
  - St. Petersburg State Government Healthcare Institution City Psychiatric Hospital #4 (St. Petersburg Insane Asylum Distributor), Saint Petersburg
- Serbia (6):
  - Institute of Mental Health, Belgrade
  - Military Medical Academy, Clinic for Psychiatry, Belgrade
  - Clinical Centre Kragujevac, Clinic for Psychiatry, Kragujevac
  - Clinical Centre Nis, Clinic for mental health protection, Niš
  - Specialized Hospital for psychiatric diseases "Sveti Vracevi", Novi Kneževac
  - Clinical Centre Vojvodina, Clinic for Psychiatry, Novi Sad
- Slovakia (7):
  - Nemonnica s poliklinikou v Prievidzi so sidlom v Bojniciach, Psychiatricke oddelenie, Bojnice
  - Psychiatricka ambulancia Mentum, s.r.o., Bratislava
  - Psychiatricka nemocnica Michalovce, Michalovce
  - PsychoLine s.r.o. Psychiatricka ambulancia, Rimavská Sobota
  - Psychiaticke oddelenie Vseobecna nemocnica Riimavska Sobota, NaP n.o., Rimavská Sobota
  - Psychiatricke oddelenie, Nemocnica s poliklinikou sv. Barbory Roznava, a.s., Rožňava
  - Centrum zdravia R. B.K. s.r.o. Psychiatricka ambulancia, Svidník
- South Africa (3):
  - Research Unit, Department of Psychiatry Free State Psychiatric Complex, Bloemfontein
  - Cape Trial Centre, Cape Town, W. Cape
  - Denmar Hospital Consulting Rooms, Pretoria

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: During the Open Label Phase subjects will receive Lurasidone 40 and 80 mg, once daily in the evening with a meal or 30 minutes after eating
- Lurasidone: During double blind phase subjects received Lurasidone flexibly dosed 40 or 80 mg once daily
- Placebo: During double blind phase subjects received matching placebo.
Period: Open Label Phase - up to 24 Weeks
Arm/Group | All Subjects | Lurasidone | Placebo
Started | 676 | 0 | 0
Completed | 287 | 0 | 0
Not Completed | 389 | 0 | 0
Not completed — Adverse Event | 83 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lack of Efficacy | 46 | 0 | 0
Not completed — Lost to Follow-up | 60 | 0 | 0
Not completed — Protocol Violation | 39 | 0 | 0
Not completed — Withdrawal by Subject | 96 | 0 | 0
Not completed — did not meet stabilization criteria | 44 | 0 | 0
Not completed — Terminated at study completion | 6 | 0 | 0
Not completed — Administrative | 14 | 0 | 0
Period: Double Blind Phase - 28 Weeks
Arm/Group | All Subjects | Lurasidone | Placebo
Started | 0 | 144 | 141
Completed | 0 | 28 | 20
Not Completed | 0 | 116 | 121
Not completed — Adverse Event | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 2 | 5
Not completed — Protocol Violation | 0 | 11 | 4
Not completed — Withdrawal by Subject | 0 | 5 | 12
Not completed — Terminated at study completion | 0 | 47 | 39
Not completed — Relapse criteria met | 0 | 43 | 58
Not completed — Administrative | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone | Placebo | Total
Number analyzed (Participants) | 144 | 141 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.38) | 42.4 (12.25) | 42.7 (11.80)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 142 | 140 | 282
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 53 | 107
  Male | 90 | 88 | 178
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 72 | 62 | 134
  White | 65 | 71 | 136
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 16
  Not Hispanic or Latino | 137 | 132 | 269
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  France | 3 | 2 | 5
  Serbia | 9 | 11 | 20
  United States | 103 | 97 | 200
  Slovakia | 11 | 11 | 22
  Russian Federation | 7 | 9 | 16
  South Africa | 10 | 11 | 21
  Italy | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to First Relapse Event During Double-blind Phase
Description: The Kaplan-Meier method is used for the estimation.
Time Frame: Double-blind phase - 28 Weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 144 | 141
days | NA [174 to NA] — Median and upper limit of the confidence interval could not be estimated. The median is not estimable for lurasidone because fewer than half of the subjects (43) had first relapse. | 192 [113 to NA] — Upper limit of the confidence interval could not be estimated.
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.039, Log Rank; Odds Ratio (OR) = 0.66, 95% CI 2-sided [0.45 to 0.98]

2. Secondary Outcome: Time to All-cause Discontinuation
Description: The Kaplan-Meier method was used for estimation.
Time Frame: Double-blind phase - 28 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 144 | 141
days | 148 [106 to NA] — Upper limit of the confidence interval could not be estimated. | 115 [82 to 148]
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.070, Log Rank; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.54 to 1.03]

3. Secondary Outcome: Change From Double-blind Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items and three scales: the Positive scale contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility; the Negative scale contains seven questions to assess blunted effect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of motivation, and similar symptoms; and the General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity.
Time Frame: Double-Blind phase - 28 Weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 144 | 141
units on a scale | 8.3 (1.33) | 12.4 (1.33)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.029, ANCOVA; LOCF

4. Secondary Outcome: Change From Double-blind Baseline in Clinical Global Impression - Severity of Illness Scale (CGI-S) Score
Description: The CGI-S score is a single value, clinician-rated assessment of illness severity and ranges from 1= 'Normal, not at all ill' to 7= 'Among the most extremely ill patients'. A higher score is associated with greater illness severity.
Time Frame: Double-blind phase - 28 Weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 144 | 141
units on a scale | 0.44 (0.087) | 0.74 (0.087)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.015, ANCOVA; LOCF

5. Secondary Outcome: Change From Double-blind Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS consists of 10 items, each rated on a Likert scale, from 0="Normal" to 6="Most Severe". The MADRS total score is calculated as the sum of the 10 items. The MADRS total score ranges from 0 to 60. Higher scores are associated with greater severity.
Time Frame: Double-blind phase - 28 Weeks
Population: There were four Lurasidone subjects and 2 placebo subjects that had no post-baseline MADRS assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 140 | 139
units on a scale | 2.5 (0.63) | 3.6 (0.63)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.218, ANCOVA; LOCF

6. Secondary Outcome: Change From Double-blind Baseline in Short Form-12v2 Health Survey (SF-12v2) Physical Component Score
Description: The SF-12v2 is a self-administered, multipurpose short-form (SF) generic measure of health status. It was developed to be a shorter, yet valid, alternative to the SF-36 for use in large surveys of general and specific populations as well as in large longitudinal studies of health outcomes. The 12 items in the SF-12v2 are a subset of those in the SF-36; SF-12v2 includes one or two items from each of the eight health concepts with higher scores indicative of higher functioning and better health. The Physical Component Score is a composite of the Physical Functioning, Role Functioning, Bodily Pain and General Health scales.
  Physical Composite Scores (PCS) is computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Double-blind phase - 28 Weeks
Population: There were 5 Lurasidone subjects and 3 placebo subjects that had no post-baseline SF-12 assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 139 | 138
units on a scale | 0.398 (0.5354) | -1.341 (0.5373)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.021, ANCOVA; LOCF

7. Secondary Outcome: Change From Double-blind Baseline in Modified Specific Levels of Functioning (SLOF) Total Score
Description: The modified SLOF scale is designed to measure directly observable behavioral functioning and daily living skills of patients with chronic mental illness. The modified SLOF consists of 24 items divided into two subscales: Social functioning (comprised of 7 items from interpersonal relationships section) and Community Living Skills (comprised of 17 items from activities and work skills sections). Each item is rated on a 5-point scale and mapped to 0 to 4 with a higher score indicating worse condition. The total score will be the sum of all 24 items and ranges from 0 to 96.
Time Frame: Double-blind phase - 28 Weeks
Population: There were 19 Lurasidone subjects and 20 placebo subjects that had no post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 125 | 121
units on a scale | 0.8 (0.88) | 3.2 (0.89)
Statistical Analysis 1: Comparison: Lurasidone vs Placebo; Test type: Superiority or Other; p = 0.056, ANCOVA; LOCF

8. Secondary Outcome: Brief Adherence Rating Scale
Description: The Brief Adherence Rating Scale (BARS) is a clinician-administered adherence assessment instrument that consists of four items including three questions and a visual analog rating scale (VAS) to assess the percentage (0 - 100%) of doses taken by the subject in the previous month.
Time Frame: Double-blind phase - 28 Weeks
Population: There were 6 Lurasidone subjects and 2 placebo subjects that had no post-baseline assessment.
Measure: Mean (Standard Deviation); unit: percentage of monthly doses taken
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 138 | 139
percentage of monthly doses taken | 98.8 (4.42) | 98.9 (3.66)

9. Other Pre Specified Outcome: EuroQol (EQ-5D): EQ-VAS Score
Description: The EQ-5D is a self-administered, standardized measure of health states consisting of two parts: EQ-5D descriptive system consisting of one question in each of five dimensions (mobility, self-care, pain, usual activities, and anxiety) with three possible response levels per question, classifying patients into one of 243 distinct health states, and a 20-cm visual analogue health status rating.
  The 20-cm visual analog scale (VAS) has endpoints labeled "best imaginable health state" and "worst imaginable health state" that are anchored at 100 and 0, respectively. Respondents are asked to indicate how they rate their own health by drawing a line from an anchor box to that point on the EQ-VAS, which best represents their own health on that day.
Time Frame: Double-blind phase - 28 Weeks
Population: There were 5 Lurasidone subjects and 3 placebo subjects that had no post-baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 139 | 138
units on a scale | 74.5 (19.87) | 68.2 (28.59)

10. Secondary Outcome: Smoking Questionnaire (Average Number of Cigarettes Per Day) at Week 28 (LOCF)
Description: Smoking history and frequency were assessed during the study by a research staff member. During the study, smoked subjects were asked about the average number of cigarettes per day they smoked over the last week.
Time Frame: 28 Weeks - Double Blind Phase
Population: ITT Subjects who smoked
Measure: Mean (Standard Deviation); unit: number of cigarettes smoked daily
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 47 | 49
number of cigarettes smoked daily | 10.0 (12.76) | 8.2 (8.97)

11. Secondary Outcome: Intent to Attend (ITA) Assessment at Open-label Baseline
Description: The ITA assessment will be administered by a research staff member. The response is recorded on a 10-point scale, with 0 = "Not at all" and 9 = "Extremely". The ITA allowed the site to capture data regarding dropout risk. The following question was completed at the screening visit: "How likely is it that you will complete the study?"
Time Frame: Open Label Baseline
Population: All subjects who were randomized and received at least one dose of study medication in the double-blind phase. Subjects were analyzed based on the treatment they were randomized.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lurasidone | Placebo
Number analyzed (Participants) | 143 | 140
units on a scale | 7.9 (1.48) | 8.0 (1.47)

ADVERSE EVENTS:
Time Frame: For the open label phase - all subjects SAEs and AEs were reported over 24 weeks. For the double blind phase, lurasidone and placebo, SAEs and AEs were reported over 28 weeks. The study was stopped once the anticipated number of relapses were reached.
Arm/Group | All Subjects | Lurasidone | Placebo
Serious Adverse Events (participants affected / at risk) | 59/676 | 6/144 | 11/141
Other Adverse Events (participants affected / at risk) | 373/676 | 46/144 | 47/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=676) | Lurasidone (N=144) | Placebo (N=141)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Artial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Drug ineffective (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Therapeutic response delayed (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponytremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Pin in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Akathasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischemic attach (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 20 (20) | 1 (1) | 4 (4)
Psychotic disorder (Psychiatric disorders) | 11 (11) | 2 (2) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hostility (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric decompensation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Substance induced psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=676) | Lurasidone (N=144) | Placebo (N=141)
Nausea (Gastrointestinal disorders) | 69 (79) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 36 (45) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 21 (31) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 22 (22) | 4 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 28 (32) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 23 (23) | 1 (1) | 1 (1)
Weight increased (Investigations) | 14 (14) | 5 (5) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 17 (21) | 6 (7) | 3 (3)
Headache (Nervous system disorders) | 77 (116) | 4 (5) | 5 (8)
Akathisia (Nervous system disorders) | 94 (104) | 3 (3) | 4 (4)
Dystonia (Nervous system disorders) | 21 (23) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 34 (38) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 24 (28) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 25 (27) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 62 (82) | 9 (10) | 10 (12)
Anxiety (Psychiatric disorders) | 35 (43) | 6 (7) | 4 (4)
Agitation (Psychiatric disorders) | 21 (22) | 3 (3) | 4 (5)
Schizophrenia (Psychiatric disorders) | 4 (4) | 10 (11) | 11 (11)
Psychotic disorder (Psychiatric disorders) | 4 (4) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In addition to the <60-180 day restriction above, since this is a multicenter study, 1st publication of study results shall be made with other participating study sites as a multicenter publication; provided, if a multicenter publication is not forthcoming within 24 months following completion of study at all sites, the PI shall be free to publish.